CLINICAL TRIAL: NCT04394325
Title: Digi-Do - a Digital Information Tool to Help Patients Diagnosed With Breast Cancer to be Involved and Prepared Before, During, and After Start of Radiotherapy Treatment
Brief Title: Digi-Do - a Digital Information Tool to Help Patients Diagnosed With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonkoping University (Other)
Responsible Party: Principal Investigator, Maria Brovall, Associate Professor, Jonkoping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: JU 2020/1732-51
Record Dates: First submitted 2020-05-06; First posted 2020-05-19 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Digital Technology; Radiotherapy (RT); Patient information; Virtual Reality (VR)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A) Intervention group (Experimental): Group A) an intervention group (n=80) who will receive the standard care and information (oral and written) + the digital information tool.
  Interventions: Behavioral: Digital information tool
- Group B) Control group (No Intervention): Group B) a control group (n=80) who will receive standard care and information (oral and written).

INTERVENTIONS:
Behavioral: Digital information tool — The patients randomized to group A will receive verbal and written information regarding the digital information tool and how to use it, as well as verbal and written information about the study. They will also receive information about the different instruments and surveys they will be asked to answer at different occasions during the RT treatment period. The applied instruments for data collection will be administrated in person or by post at the baseline collection and by post (including pre-paid return envelope) on consecutive collections. Approximately 30 patients (in group A) will be asked to make regular notes in a notebook during the waiting period prior start of RT as well as during RT treatment period. Following completion of the RT treatment period individual in-depth and telephone interviews will take place with 10-12 patients that accept participation.
  Arms: Group A) Intervention group

SUMMARY:
This project uses participatory design combined with qualitative and quantitative methods to develop, explore and evaluate the usefulness of a digital information tool to prepare and support patients before, during and after RT as treatment for breast cancer.

DETAILED DESCRIPTION:
The study is a prospective and longitudinal Randomised Control Trial (RCT) study with an Action Research (AR) participatory design approach, including mixed-method data collection, i.e., standardised instruments, interviews (face-to-face and telephone), diaries, observation, and time measurements. The timeline for the study is scheduled between autumn 2020 to spring 2022. The study will consist of two arms: A) an intervention group (n=80), who will receive standard care and information and the digital information tool; and B) a control group (n=80) who will receive standard care and information (verbal and written). Recruitment and randomisation will be completed at two hospitals in the South western part of Sweden.

As a pre-phase, a pilot study was performed for the development and testing of the digital information tool (Digi-Do), approved by the Regional Ethics Committee (Dnr 917-17) with 30 patients in total (15 women with breast cancer and 15 men with prostate cancer). According to the study's co-design, iterative methodology [26-27 in manuscript], changes have since been made to the digital information tool and a second version has now been developed for the full RCT. The present study has been approved by the Swedish Ethical Review Authority (Dnr 2020-00170). An ongoing systematic literature review will also guide the present study, and the project is registered in PROSPERO (PROSPERO;168073).

The digital information tool applied in this project is divided into two separate but coherent applications (apps) for mobile devices: one (VR-app) with a guided tour of the RT-department with a voice-over to describe 360 images to create a sense of actually having visited the department prior to start of RT, and one (information app) containing information obtained through the pre-treatment phase. If a VR-effect is not desirable, the patient can complete the simulated study-visit on their mobile phone or tablet as well as present the images in the browser of an integrated media player. Three areas of information are available in the information app: 1) Q&As from the existing written information, presented both in writing and a recorded voice; 2) practical information, such as maps, public transportation options with relevant links to public transport, telephone numbers, and information about possibilities for staying at the patient hotel; and 3) three short animated films about cancer and physical activity during RT.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (>18 years):

* diagnosed with breast cancer, stage I-II not receiving adjuvant or neo-adjuvant chemotherapy or anti-Her-2 treatment and
* with RT as additional treatment after surgery.
* ability to read, write and understand Swedish enough to adhere to the digital information tool and the applied instruments.
* that have access to a smartphone.

Exclusion Criteria:

* not receiving RT have had RT before
* diagnosed with dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change in distress | Baseline pre intervention
  The National Comprehensive Cancer Network Distress Thermometer is a brief screening tool for cancer patients to assess psychosocial distress
Change in distress | up to one week of intervention
  The National Comprehensive Cancer Network Distress Thermometer is a brief screening tool for cancer patients to assess psychosocial distress
Change in distress | 6 months after the intervention
  The National Comprehensive Cancer Network Distress Thermometer is a brief screening tool for cancer patients to assess psychosocial distress

SECONDARY OUTCOMES:
Change in general self-efficacy | Baseline pre intervention
  The Swedish version of the General Self-efficacy (GSE) Scale. The GSE scale consists of 10 items rated on a fourpoint Likert scale (''not at all true'' to ''exactly true'').
Change in general self-efficacy | 6 months after the intervention
  The Swedish version of the General Self-efficacy (GSE) Scale. The GSE scale consists of 10 items rated on a fourpoint Likert scale (''not at all true'' to ''exactly true'').
Change in communicative and critical health literacy | Baseline pre intervention
  The communicative and critical health literacy scale - Swedish version. The first three items include statements focusing on the capacity for collecting, extracting, and understanding relevant health information. Each item is rated on a 4-point scale, ranging from 1 (never=better) to 4 (often=worse).
Change in communicative and critical health literacy | 6 months after the intervention
  The communicative and critical health literacy scale - Swedish version. The first three items include statements focusing on the capacity for collecting, extracting, and understanding relevant health information. Each item is rated on a 4-point scale, ranging from 1 (never=better) to 4 (often=worse).
Change in functional health literacy | Baseline pre intervention
  The Swedish Functional Health Literacy scale scale comprises five items about persons' skills in reading and understanding health information. Each item is rated on a 4-point scale, ranging from 1 (never=better) to 4 (often=worse).
Change in functional health literacy | 6 months after the intervention
  The Swedish Functional Health Literacy scale scale comprises five items about persons' skills in reading and understanding health information. Each item is rated on a 4-point scale, ranging from 1 (never=better) to 4 (often=worse).
Change in eHealth literacy | Baseline pre intervention
  The The eHealth Literacy Questionnaire (eHLQ) is a psychometrically robust multidimensional tool designed to be used to understand and evaluate people's interaction with digital health services
Change in eHealth literacy | 6 months after the intervention
  The The eHealth Literacy Questionnaire (eHLQ) is a psychometrically robust multidimensional tool designed to be used to understand and evaluate people's interaction with digital health services
Time measurements and Observations | up to one week of intervention
  Ten patients respectively from groups A and B will be consequently asked to participate in the time measurement and observational part of the study (n=20). All planned treatments for the first week of RT (n=5), and, additionally, one session in the last week of treatment, will be measured based on seven timepoints; patient enters door of RT room, patient lies on table, first image, first field beam on, last field beam on, patient leaves table, and patient leaves RT room. This will result in approximately 120 points of measurement. During each RT session, observations of questions asked by patients and staff will be documented in a protocol, including what subjects are addressed, who initiates the question, and whether, how, and to where the staff refers the patient for further information.
Time measurements and Observations | up to five week of intervention
  Ten patients respectively from groups A and B will be consequently asked to participate in the time measurement and observational part of the study (n=20). All planned treatments for the first week of RT (n=5), and, additionally, one session in the last week of treatment, will be measured based on seven timepoints; patient enters door of RT room, patient lies on table, first image, first field beam on, last field beam on, patient leaves table, and patient leaves RT room. This will result in approximately 120 points of measurement. During each RT session, observations of questions asked by patients and staff will be documented in a protocol, including what subjects are addressed, who initiates the question, and whether, how, and to where the staff refers the patient for further information.

OTHER OUTCOMES:
In-depth interviews | 1 week after the intervention
  The individual in-depth and/or telephone interviews will take place on two occasions (1-4 weeks and 6 months post-RT completion) and with at least ten of the patients who have accepted participation and have made regular notes. Questions will include topics such as their experiences of receiving the information through the digital information tool during the waiting time and treatment period, of using the digital information tool, to what extent the digital information has affected their involvement and preparedness for the radiation treatment, as well as their experiences during the time since the end of RT
In-depth interviews | 6 months after the intervention
  The individual in-depth and/or telephone interviews will take place on two occasions (1-4 weeks and 6 months post-RT completion) and with at least ten of the patients who have accepted participation and have made regular notes. Questions will include topics such as their experiences of receiving the information through the digital information tool during the waiting time and treatment period, of using the digital information tool, to what extent the digital information has affected their involvement and preparedness for the radiation treatment, as well as their experiences during the time since the end of RT

CONTACTS AND LOCATIONS:
Overall Officials: maria brovall, Principal Investigator — Jonkoping Univeristy Box 1026, 551 11 Jonkoping
Locations (1):
- Sahlgrenska universitetssjukhuset, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fristedt S, Smith F, Grynne A, Browall M. Digi-Do: a digital information tool to support patients with breast cancer before, during, and after start of radiotherapy treatment: an RCT study protocol. BMC Med Inform Decis Mak. 2021 Feb 25;21(1):76. doi: 10.1186/s12911-021-01448-3. PMID 33632215